CLINICAL TRIAL: NCT06060730
Title: Translation, Cultural Adaptation, Reliability, and Validity of the Turkish Version of the Patellofemoral Pain and Osteoarthritis Subscale of the KOOS (KOOS PF)
Brief Title: Measurement Properties of the Turkish Version of the Patellofemoral Pain and Osteoarthritis Subscale of the KOOS
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sevim Beyza Ölmez, Principal investigator, Gazi University
Other Study IDs: 2023 - 986
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Patellofemoral Pain Syndrome; Patellofemoral Osteoarthritis; PROMs
Keywords: Patellofemoral Pain Syndrome; Patellofemoral Osteoarthritis; Patient-reported outcome measures; PROMs; Validity; Reliability
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to translate and culturally adapt the subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) into Turkish, and to determine the measurement properties of the Turkish version.

DETAILED DESCRIPTION:
Patellofemoral pain and patellofemoral osteoarthritis are highly prevalent knee disorders associated with pain and functional limitations. Patient-reported outcome measures (PROMs) are suggested for clinical and research use; however, there is a lack of objective disease-specific PROMs for patellofemoral pain and osteoarthritis. The purpose of this study is to translate and culturally adapt the subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) into Turkish, and to determine the measurement properties of the Turkish version.

ELIGIBILITY:
Inclusion Criteria:

* peripatellar or retropatellar knee pain persisting for at least 3 months and exacerbated by activities that load the patellofemoral joint;
* pain intensity of at least 3 mm according to the visual analogue scale (VAS)

Exclusion Criteria:

* diffuse or generalized knee pain
* severe trauma to the target knee in the previous year
* moderate to severe concomitant tibiofemoral osteoarthritis
* recent knee injection (within 3 months)
* systemic inflammatory conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with patellofemoral pain and OA
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
the subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) | first day
  The subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) is a disease-specific PROM designed to evaluate pain, stiffness, and quality of life in patients with patellofemoral pain and/or osteoarthritis. It has 11 items that assess three domains: stiffness (1 item), pain (9 items), and quality of life (1 item). Each item consists of five response options with a score between 0 and 4. The total score ranges from 0 (worst) to 100 (best).
the Kujala's Anterior Pain Scale (AKPS) | first day
  The Kujala's Anterior Pain Scale (AKPS) is a self-administered questionnaire designed for patellofemoral disorders. It consists of 13 items on symptoms and functional limitations. The total score ranges from 0 to 100, with higher values indicating less functional status
the Short Form-36 health survey (SF-36) | first day
  The short-form 36 (SF-36) health survey is a tool for assessing general health-related quality of life. It consists of 36 questions divided into eight domains, which are then merged under two large headings: physical component summary and mental component summary. The total score varies between 0 and 100. Higher ratings indicate a better quality of life.
the subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) | 7-14 days after
  The subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) is a disease-specific PROM designed to evaluate pain, stiffness, and quality of life in patients with patellofemoral pain and/or osteoarthritis. It has 11 items that assess three domains: stiffness (1 item), pain (9 items), and quality of life (1 item). Each item consists of five response options with a score between 0 and 4. The total score ranges from 0 (worst) to 100 (best).
the subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) | 3 months after
  The subscale of the Knee Injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) is a disease-specific PROM designed to evaluate pain, stiffness, and quality of life in patients with patellofemoral pain and/or osteoarthritis. It has 11 items that assess three domains: stiffness (1 item), pain (9 items), and quality of life (1 item). Each item consists of five response options with a score between 0 and 4. The total score ranges from 0 (worst) to 100 (best).
the global rating of change (GROC) | 3 months after
  The global rating of change (GROC) score is a single-item questionnaire with five potential responses depending on the patient's change in knee pain following the initial assessment. Likert scale with five response options: "0 points" (much worse), "1 points" (slightly worse), "2 points" (about the same), "3 points" (slightly better), and "4 points" (much better).

CONTACTS AND LOCATIONS:
Overall Officials: Selda Başar, Prof, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)